CLINICAL TRIAL: NCT06578572
Title: Seasonal R21 Mass Vaccination for Malaria Elimination
Acronym: SERVAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Malaria Control Programme, The Gambia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LEO29834
Record Dates: First submitted 2024-03-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Malaria
Keywords: Malaria; Malaria vaccine R21/Matrix M; Mass vaccination; The Gambia; Burkina Faso
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Three monthly doses of R21/MM will be administered to all eligible residents in the 27 intervention villages (15 in The Gambia and 12 in Burkina Faso), starting from May 2024, with the aim of having completed the vaccination schedule by end of July 2024, before the malaria transmission season starts. A booster vaccine dose will be administered in June 2025 to all eligible individuals who received at least one vaccine dose the previous year. Residents who are eligible but not vaccinated in the previous year, will be offered a complete vaccination schedule, i.e. 3 monthly doses, starting from April. After each vaccination, the first 100 vaccinated individuals will be visited at home daily, for 3 consecutive days, and then at day 7 after the vaccination to collect local and systemic adverse events (AE). Vaccinated individuals (or their parents) will be asked to report to the nurse based in their study village any illness occurring during the 28 days after vaccination.
  Interventions: Biological: R21Matrix M
- Control Group (No Intervention): Only standard malaria control measures ( Malaria Chemoprevention (SMC), Intermittent Preventive Treatment during pregnancy (IPTp), Insecticide-Treated bed Nets (ITN), prompt diagnosis and treatment of patients with uncomplicated malaria and Indoor Residual Spraying (IRS)) will be implemented in control villages.

INTERVENTIONS:
Biological: R21Matrix M — A mixture of R21/Matrix M at a dose of 5 μg (for children up to 14 years of age) or 10 μg ( for individuals ≥ 15 years old) with 50 μg of Matrix-M will be administered monthly over 3 months (one dose per month over 3 months (May, June, and July 2024) plus a booster dose in June 2025.
  Arms: Experimental Group

SUMMARY:
This is a cluster randomized trial to determine the impact of seasonal R21/MM mass vaccination (all ages) on malaria transmission and morbidity. Fifty-four villages (30 in The Gambia and 24 in Burkina Faso) will be randomized to either mass vaccination with R21 or no mass vaccination.

The primary objective is to compare in intervention and control clusters the prevalence of malaria (all age groups) at peak transmission after seasonal mass vaccination with R21 (3 monthly doses).

Secondary objectives are:

1. To assess the safety and tolerability of R21 through spontaneously reported adverse events.
2. To compare in intervention and control clusters the incidence of malaria infection (all age groups) during the malaria transmission season following seasonal mass vaccination with R21 (3 monthly doses).
3. To compare in intervention and control clusters the incidence of clinical malaria (all age groups) after seasonal mass vaccination with R21 (3 monthly doses).
4. To compare in intervention and control clusters the prevalence of malaria (all age groups) at peak transmission after one booster dose of R21.
5. To compare in intervention and control clusters the incidence of malaria infection (all age groups) during the malaria transmission season following one booster dose of R21.
6. To compare in intervention and control clusters the incidence of clinical malaria (all age groups), after one booster dose of R21.
7. To determine the coverage of seasonal mass vaccination with R21 (primary series of three vaccinations and booster) in intervention clusters and related socio-cultural factors
8. To estimate the cost of seasonal mass vaccination with R21 administration.
9. To estimate the cost-effectiveness of seasonal mass vaccination with R21 compared to standard malaria control measures.

The exploratory objective is to determine whether serological markers can detect changes in malaria transmission following mass vaccination with R21.

DETAILED DESCRIPTION:
This is a cluster-randomized controlled trial. Fifty-four villages (30 in The Gambia and 24 in Burkina Faso) will be randomized to either mass vaccination with R21 or no mass vaccination. Therefore,15 medium-sized (200-600 people) villages in The Gambia and 12 medium-sized (200-600 people) villages in Burkina Faso will receive the intervention. All study villages will receive standard control intervention, e.g., seasonal malaria chemoprevention, insecticide-treated bed nets, implemented by the National Malaria Control Program and according the National Strategic Plan for malaria control. Mass vaccination will be completed before the start of the malaria transmission season, i.e. July.

A cross-sectional survey to estimate malaria prevalence will be implemented at peak transmission, both following the mass vaccination with 3 doses (first year) and the booster dose (second year). A blood sample will be collected during the malaria transmission season from a cohort of randomly selected individuals to determine the incidence of malaria infection. A system of passive case detection to determine the incidence of clinical malaria will be set up throughout the study period, with special attention to the malaria transmission season (July-December).

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 5 months.
2. Willingness to comply with trial procedures.
3. Individual written informed consent obtained at the beginning of the study.

Exclusion Criteria:

1. Pregnancy
2. History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g., Kathon, neomycin, betapropiolactone.
3. Any history of anaphylaxis in relation to vaccination.
4. Known chronic illness.
5. Any other significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 5 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16200 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malaria infection by PCR in all age groups at peak transmission season (October-November) following the first vaccination with 3 doses. | At 6 months ( October - November 2024) post first round of vaccination
  A cross-sectional survey will be conducted at peak transmission in October -November 2024 to determine prevalence of malaria infection.

SECONDARY OUTCOMES:
Occurrence of Adverse Events (AEs) during follow up. | Up to 28 days post vaccination
  1. Occurrence of solicited local and/or systemic reactogenicity
  2. Occurrence of unsolicited adverse events
  3. Occurrence of abnormal hematology and biochemistry parameters ( clinically significant values)
  4. Occurrence of serious adverse events ( throughout the trial)
Incidence of malaria infection in all age groups during the transmission season following mass vaccination with R21 | Up to 6 months post the third vaccination round
  Incidence of malaria infection will be determined by molecular analyses (PCR) in a cohort of 20 individuals per village in Burkina Faso and 30 individuals per villages in The Gambia through monthly home visits ( following mass vaccination with R21).
Incidence of clinical malaria in all age groups following mass vaccination with R21. | Up to 6 months post the third vaccination round
  A passive case detection of clinical malaria throughout the study period, with special attention to the malaria transmission season (July-December)
Prevalence of malaria infection by PCR in all age groups at peak transmission following the booster dose. | At 6 months ( October - November 2025) post booster dose
  A cross-sectional survey will be conducted at peak transmission in October -November 2025 to determine prevalence of malaria infection.
Incidence of malaria infection in all age groups during the transmission season following the booster dose. | Up to 6 months post booster dose
  Incidence of malaria infection will be determined by molecular analyses (PCR) in a cohort of 20 individuals per village in Burkina Faso and 30 individuals per villages in The Gambia through monthly home visits ( following the booster dose).
Incidence of clinical malaria in all age groups following the booster dose. | Up to 6 months post the third vaccination round
  Passive detection of clinical malaria both at the community and at health facility level
Coverage of completed vaccination schedule (3 doses) during the mass vaccination with 3 doses. | Up to 4 weeks post the third vaccination round
  Coverage of completed vaccination schedule (3 doses) during the mass vaccination with 3 doses.
Coverage of at least one vaccine dose administered during the mass vaccination with 3 doses | Up to 4 weeks post the third vaccination round
  Coverage of at least one vaccine dose
Coverage of the booster dose | Up to 4 weeks post booster dose
  Coverage of the booster dose
Cost of vaccine administration and cost effectiveness, both for the mass vaccination campaign with 3 doses and the booster dose. | Up to 6 months post booster dose
  A cross sectional survey will be carried out at the beginning of the project in both study arms to estimate the cost of seeking care among households and the costs supported by the health facility. Cost of mass vaccination will be collected for each round.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD, MSc, PhD, Principal Investigator — MRCG at LSHTM; Halidou Tinto, PhD, Principal Investigator — Clinical Research Unit of Nanoro (CRUN); Edgard Dabira, MD, MSc, PhD, Study Director — MRCG at LSHTM; Magloire Natama, PhD, Study Director — Clinical Research Unit of Nanoro, Burkina Faso
Locations (2):
- Clinical Research Unit of Nanoro, Burkina Faso, Nanoro, Burkina Faso
- MRC Unit The Gambia at LSHTM, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD data will be made available from one month after trial publication and for a further 24 months
Supporting Information: Study Protocol, ICF
Time Frame: 1 month after the publication date and for a further 24 months
Access Criteria: Application to the principal investigator with a justification of the request

REFERENCES:
- [Derived] Dabira ED, Natama HM, Jaiteh F, Grietens KP, Bocoum FY, Ndiath MO, Mohammed N, Gibba B, Hill AVS, Ghani A, Erhart A, Tinto H, D'Alessandro U. Seasonal mass vaccination with R21/Matrix-M for malaria elimination (SERVAL): protocol of the cluster randomised trial. Trials. 2025 Sep 29;26(1):382. doi: 10.1186/s13063-025-09048-6. PMID 41024138